CLINICAL TRIAL: NCT01799941
Title: A Study to Assess the Safety, Tolerability and Effectiveness of Nuedexta (Dextromethorphan 20 mg/Quinidine 10 mg) in the Treatment of Pseudobulbar Affect (PBA)
Brief Title: Safety, Tolerability and Effectiveness of Nuedexta in the Treatment of Pseudobulbar Affect (PBA)
Acronym: PRISM II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-AVR-401
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Pseudobulbar Affect (PBA); Stroke; Dementia; Traumatic Brain Injury (TBI)
MeSH Terms: conditions — Stroke; Dementia; Brain Injuries, Traumatic | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nuedexta (DM 20 mg/Q 10 mg) (Other): Single Arm, Open Label Dosing with Nuedexta (DM 20 mg/Q 10 mg)
  Interventions: Drug: Nuedexta (DM 20 mg/Q 10 mg)

INTERVENTIONS:
Drug: Nuedexta (DM 20 mg/Q 10 mg) — Single Arm, Open-Label Dosing with Nuedexta (DM 20 mg/Q 10 mg)
  Other Names: Nuedexta

SUMMARY:
The objectives of the study are to evaluate the safety, tolerability, and effectiveness of NUEDEXTA capsules containing 20 mg DM (Dextromethorphan)/10 mg Q (Quinidine) for treatment of Pseudobulbar Affect (PBA) in patients with prevalent conditions such as dementia, stroke, and traumatic brain injury (TBI)over a 12 week period.

DETAILED DESCRIPTION:
This will be an Open-label, Multicenter, study in patients with PBA and dementia, stroke or TBI. Patients with a clinical diagnosis of PBA and who meet all other inclusion and exclusion criteria will be eligible to participate and receive NUEDEXTA for 12 weeks.

Males and females patients with a minimum age of 18 years, a clinical diagnosis of Pseudobulbar Affect and a documented diagnosis of neurologic disease or brain injury, will be enrolled in this study.

The primary effectiveness endpoint is the mean change in the Center for Neurologic Study-Lability scale (CNS-LS). Secondary objectives include measures to evaluate treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Center for Neurologic Study-Lability Scale (CNS-LS)score of 13 or greater
* Clinical diagnosis of Pseudobulbar Affect (PBA)
* Documentation of Neurologic disease or brain injury

Exclusion Criteria:

* Unstable neurologic disease
* Severe dementia
* Stroke within 3 months
* Penetrating TBI
* Contraindications to Nuedexta
* Severe Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pensacola, Florida, United States

REFERENCES:
- [Derived] Hammond FM, Sauve W, Ledon F, Davis C, Formella AE. Safety, Tolerability, and Effectiveness of Dextromethorphan/Quinidine for Pseudobulbar Affect Among Study Participants With Traumatic Brain Injury: Results From the PRISM-II Open Label Study. PM R. 2018 Oct;10(10):993-1003. doi: 10.1016/j.pmrj.2018.02.010. Epub 2018 Feb 23. PMID 29477412
- [Derived] Hammond FM, Alexander DN, Cutler AJ, D'Amico S, Doody RS, Sauve W, Zorowitz RD, Davis CS, Shin P, Ledon F, Yonan C, Formella AE, Siffert J. PRISM II: an open-label study to assess effectiveness of dextromethorphan/quinidine for pseudobulbar affect in patients with dementia, stroke or traumatic brain injury. BMC Neurol. 2016 Jun 9;16:89. doi: 10.1186/s12883-016-0609-0. PMID 27276999
- [Derived] Doody RS, D'Amico S, Cutler AJ, Davis CS, Shin P, Ledon F, Yonan C, Siffert J. An open-label study to assess safety, tolerability, and effectiveness of dextromethorphan/quinidine for pseudobulbar affect in dementia: PRISM II results. CNS Spectr. 2016 Dec;21(6):450-459. doi: 10.1017/S1092852915000620. Epub 2015 Oct 16. PMID 26471212

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 394 participants were screened of which 367 participants were enrolled in the study; 134 in the dementia cohort, 113 in the stroke cohort, and 120 in the traumatic brain injury (TBI) cohort.
Groups:
- Dextromethorphan Hydrobromide 20 mg + Quinidine Sulfate 10 mg: Participants who received fixed-dose combination of 20 milligram (mg) dextromethorphan hydrobromide and 10 mg quinidine sulfate, orally once daily in the morning for the first week of the study, and twice daily (every 12 hours) for the remaining 11 weeks of the study.
Period: Overall Study
Arm/Group | Dextromethorphan Hydrobromide 20 mg + Quinidine Sulfate 10 mg
Started | 367
Completed | 271
Not Completed | 96
Not completed — Adverse Event | 34
Not completed — Withdrawal by Subject | 21
Not completed — Death | 2
Not completed — Investigator Decision | 4
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 17
Not completed — Other | 15

BASELINE CHARACTERISTICS:
Groups:
- Dextromethorphan Hydrobromide 20 mg + Quinidine Sulfate 10 mg: Participants who received fixed-dose combination of 20 mg dextromethorphan hydrobromide and 10 mg quinidine sulfate, orally once daily in the morning for the first week of the study, and twice daily (every 12 hours) for the remaining 11 weeks of the study.
Arm/Group | Dextromethorphan Hydrobromide 20 mg + Quinidine Sulfate 10 mg
Number analyzed (Participants) | 367
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 215
  >=65 years | 152
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 165

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Center for Neurologic Study-Lability Scale (CNS-LS) Score at Day 90
Description: The CNS-LS was a seven-item, self-administered questionnaire, completed by the participant or participant's caregiver that provided a quantitative measure of the perceived frequency and severity of Pseudobulbar Affect (PBA) episodes. It consisted of two subscales measuring labile laughter (four items) and labile crying (three items). Each item was rated on a scale from 1 (applies never) to 5 (applies most of the time). The total score was calculated as the sum of the item values that resulted in a score ranging from 7 (no symptoms) to 35 (maximum symptom severity and frequency). A single continuous variable was created for the reported time point. The change in CNS-LS was calculated as the score from the Day 90 assessment minus the Baseline CNS-LS measure. A negative change represented a decrease in CNS-LS score over time following the baseline assessment indicating a perceived decrease in frequency and severity of PBA episodes.
Time Frame: Day 90 (Final visit)
Population: The analysis was performed using the Modified Intent-to-treat (mITT) Population, defined as all participants who met all inclusion criteria, with a score of at least 13 on the CNS-LS, who received at least 1 dose of study drug, and who had at least 1 post-baseline efficacy measurement with CNS-LS.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Overall: Participants with dementia, stroke, and traumatic brain injury who received fixed-dose combination of 20 mg dextromethorphan hydrobromide and 10 mg quinidine sulfate, orally once daily in the morning for the first week of the study, and twice daily (every 12 hours) for the remaining 11 weeks of the study.
- Dementia: Participants with dementia who received fixed-dose combination of 20 mg dextromethorphan hydrobromide and 10 mg quinidine sulfate, orally once daily in the morning for the first week of the study, and twice daily (every 12 hours) for the remaining 11 weeks of the study.
- Stroke: Participants with stroke who received fixed-dose combination of 20 mg dextromethorphan hydrobromide and 10 mg quinidine sulfate, orally once daily in the morning for the first week of the study, and twice daily (every 12 hours) for the remaining 11 weeks of the study.
- Traumatic Brain Injury: Participants with traumatic brain injury who received fixed-dose combination of 20 mg dextromethorphan hydrobromide and 10 mg quinidine sulfate, orally once daily in the morning for the first week of the study, and twice daily (every 12 hours) for the remaining 11 weeks of the study.
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 261 | 102 | 92 | 67
Units on a scale | -7.69 (6.07) | -7.22 (6.04) | -7.59 (6.67) | -8.54 (5.18)
Statistical Analysis 1: Comparison: Overall; The primary analysis tested the null hypothesis that the mean change in CNS-LS score from Baseline to Day 90 visit is equal to zero; Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 2: Comparison: Dementia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, one-sample t-test
Statistical Analysis 3: Comparison: Stroke; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 4: Comparison: Traumatic Brain Injury; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 5: Comparison: Dementia vs Stroke; Test type: Superiority or Other; Analysis of covariance (ANCOVA) = 0.04, 95% CI 2-sided [-1.37 to 1.45], Standard Error of Mean 0.72 — A positive estimate indicates a smaller change in the first group. Observations used =261
Statistical Analysis 6: Comparison: Stroke vs Traumatic Brain Injury; Test type: Superiority or Other; ANCOVA = 1.11, 95% CI 2-sided [-0.46 to 2.68], Standard Error of Mean 0.80 — A positive estimate indicates a smaller change in the first group. Observations used =261
Statistical Analysis 7: Comparison: Dementia vs Traumatic Brain Injury; Test type: Superiority or Other; ANCOVA = 1.15, 95% CI 2-sided [-0.39 to 2.69], Standard Error of Mean 0.78 — A positive estimate indicates a smaller change in the first group. Observations used =261

2. Secondary Outcome: Mean Change From Baseline in Center for Neurologic Study-Lability Scale (CNS-LS) Score at Day 30
Description: The CNS-LS was a seven-item, self-administered questionnaire, completed by the participant or participant's caregiver that provided a quantitative measure of the perceived frequency and severity of Pseudobulbar Affect (PBA) episodes. It consisted of two subscales measuring labile laughter (four items) and labile crying (three items). Each item was rated on a scale from 1 (applies never) to 5 (applies most of the time). The total score was calculated as the sum of the item values that resulted in a score ranging from 7 (no symptoms) to 35 (maximum symptom severity and frequency). A single continuous variable was created for the reported time point. The change in CNS-LS was calculated as the score from the Day 30 assessment minus the Baseline CNS-LS measure. A negative change represented a decrease in CNS-LS score over time following the baseline assessment indicating a perceived decrease in frequency and severity of PBA episodes.
Time Frame: Day 30
Population: The analysis was performed using the mITT population, defined as all participants who met all inclusion criteria, with a score of at least 13 on the CNS-LS, who received at least 1 dose of study drug, and who had at least 1 post-baseline efficacy measurement with CNS-LS.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 297 | 108 | 103 | 86
Units on a scale | -5.43 (5.52) | -4.60 (5.08) | -6.17 (6.12) | -5.58 (5.21)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 2: Comparison: Dementia; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 3: Comparison: Stroke; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 4: Comparison: Traumatic Brain Injury; Test type: Superiority or Other; p < 0.0001, One-sample t-test

3. Secondary Outcome: Mean Pseudobulbar Affect (PBA) Episode Count Per Week by Visit
Description: PBA episode count was an investigator assessed measure in which the participant/participant's daytime caregiver was asked to identify, count and recall the total episodes of exaggerated/uncontrollable laughing or crying over the previous 7 days (prior to visit) at Baseline (Day 1), Day 30 (Visit 1), and Day 90 (Final visit). The response categories for this question were: 0, 1- 2, 3-5, 6-10, >10. The original responses from participants were converted to estimate the continuous number of PBA episodes by taking the mid-point of the original response ranges and multiplying that value by 7. Data is presented as mean PBA count per week.
Time Frame: Baseline (Day 1), Day 30 (Visit 1), and Day 90 (Final visit)
Population: The analysis population consisted of all participants who met all inclusion criteria, including a score of at least 13 on the CNS-LS, who received at least 1 dose of study drug, and who had at least 1 post-baseline efficacy measurement with PBA episode.
Measure: Mean (Standard Deviation); unit: Count/week
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 298 | 108 | 103 | 87
Count/week
  Baseline | 21.33 (24.97) | 25.68 (23.06) | 19.62 (29.62) | 17.94 (20.31)
  Day 30 (n= 296, 108, 102, 86) | 9.10 (14.29) | 12.85 (16.80) | 6.95 (11.83) | 6.94 (12.60)
  Day 90 (n= 260, 102, 92, 66) | 6.23 (11.45) | 8.41 (14.26) | 5.26 (9.60) | 4.20 (8.02)
Statistical Analysis 1: Comparison: Overall; Day 30 versus Baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 2: Comparison: Overall; Day 90 versus Baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 3: Comparison: Dementia; Day 30 versus Baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 4: Comparison: Dementia; Day 90 assessment; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 5: Comparison: Stroke; Day 30 versus Baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 6: Comparison: Stroke; Day 90 versus Baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 7: Comparison: Traumatic Brain Injury; Day 30 versus Baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 8: Comparison: Traumatic Brain Injury; Day 90 versus Baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test

4. Secondary Outcome: Percentage of Participants With PBA Remission
Description: PBA remission was defined as participants with one or more episodes reported at the baseline (Day 1) visit and zero episodes reported at the Day 30 (Visit 1) or Day 90 (Final visit). Data is reported as percentage of participants with no reported episodes over the previous 7 days (prior to visit) at Day 30 (Visit 1) and Day 90 (Final visit).
Time Frame: Day 30 (Visit 1) and Day 90 (Final visit)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 298 | 108 | 103 | 87
Percentage of participants
  Day 30 (n= 296, 108, 102, 86) | 20.3 | 13.0 | 22.5 | 26.7
  Day 90 (n= 260, 102, 92, 66) | 35.4 | 31.4 | 34.8 | 42.4

5. Secondary Outcome: Percentage Change From Baseline in PBA Episode Count Per Week
Description: The change from the baseline PBA rate was measured using Mixed Effects Poisson Regression Model (adjusted for gender and age [≤ 65 years]).
Time Frame: Day 30 (Visit 1) and Day 90 (Final visit)
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 298 | 108 | 103 | 87
percent change
  Day 30 (n= 296, 108, 102, 86) | -57.5 [-59.3 to -55.5] | -50.0 [-53.1 to -46.6] | -64.9 [-67.7 to -61.7] | -61.3 [-64.8 to -57.7]
  Day 90 (n=260, 102, 92, 66) | -72.3 [-73.8 to -70.8] | -67.7 [-70.1 to -65.1] | -74.5 [-76.9 to -71.8] | -78.5 [-81.2 to -75.7]
Statistical Analysis 1: Comparison: Overall; Day 30 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regreesion Model; Incidence Rate Ratio = 0.425, 95% CI 2-sided [0.407 to 0.445], Standard Error of Mean 0.023 — Number of observations = 854, Number of participants = 298
Statistical Analysis 2: Comparison: Overall; Day 90 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regression Model; Incidence Rate Ratio = 0.277, 95% CI 2-sided [0.262 to 0.293], Standard Error of Mean 0.028 — Number of observations = 854, Number of participants = 298
Statistical Analysis 3: Comparison: Dementia; Day 30 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regression Model; Incidence Rate Ratio = 0.500, 95% CI 2-sided [0.469 to 0.534], Standard Error of Mean 0.033 — Number of observations = 318, Number of participants = 108
Statistical Analysis 4: Comparison: Dementia; Day 90 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regression Model; Incidence Rate Ratio = 0.323, 95% CI 2-sided [0.299 to 0.349], Standard Error of Mean 0.039 — Number of observations = 318, Number of participants = 108
Statistical Analysis 5: Comparison: Stroke; Day 30 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regression Model; Incidence Rate Ratio = 0.351, 95% CI 2-sided [0.323 to 0.383], Standard Error of Mean 0.044 — Number of observations = 297, Number of participants = 103
Statistical Analysis 6: Comparison: Stroke; Day 90 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regression Model; Incidence Rate Ratio = 0.255, 95% CI 2-sided [0.231 to 0.282], Standard Error of Mean 0.051 — Number of observations = 297, Number of participants = 103
Statistical Analysis 7: Comparison: Traumatic Brain Injury; Day 30 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regression Model; Incidence Rate Ratio = 0.387, 95% CI 2-sided [0.352 to 0.425], Standard Error of Mean 0.048 — Number of observations = 239, Number of participants = 87
Statistical Analysis 8: Comparison: Traumatic Brain Injury; Day 90 assessment; Test type: Superiority or Other; p < 0.0001, Mixed Effects Poisson Regression Model; Incidence Rate Ratio = 0.215, 95% CI 2-sided [0.189 to 0.245], Standard Error of Mean 0.066 — Number of observations = 239, Number of participants = 87

6. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction in PBA Episode Count Per Week
Description: Data is reported as the percentage of participants with ≥ 50% reduction in PBA episode count/week.
Time Frame: Day 30 (Visit 1) and Day 90 (Final visit)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 298 | 108 | 103 | 87
Percentage of participants
  Day 30 (n= 289, 107, 100, 82) | 63.7 | 58.9 | 65.0 | 68.3
  Day 90 (n= 254, 101, 90, 63) | 78.0 | 76.2 | 76.7 | 82.5

7. Secondary Outcome: Percentage of Participants With ≥ 75% Reduction in PBA Episode Count Per Week
Description: Data is reported as the percentage of participants with ≥ 75% reduction in PBA episode count/week.
Time Frame: Day 30 (Visit 1) and Day 90 (Final visit)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 298 | 108 | 103 | 87
Percentage of participants
  Day 30 (n= 289, 107, 100, 82) | 42.2 | 33.6 | 42.0 | 53.7
  Day 90 (n= 254, 101, 90, 63) | 57.1 | 57.4 | 47.8 | 69.8

8. Secondary Outcome: Mean Change From Baseline in Quality of Life Visual Analog Scale (QOL-VAS) Score at Day 90
Description: The QOL-VAS, a participant reported scale of quality of life (QOL) was used to measure the impact of PBA episodes on the participant's QOL over the previous 7 days (prior to visit) at Baseline (Day 1) and Day 90 (Final visit). The assessment was completed by a participant placing a mark on a horizontal line that extends from 0 "not (affected) at all" to 10 "significantly (affected)". The participant's mark was measured and recorded at each time point. The change in QOL-VAS score from baseline to day 90 visit, defined as the day 90 score minus the baseline score, was analyzed. Data is reported as mean QOL-VAS score; a positive change in score represented an increase in participant's quality of life.
Time Frame: Day 90 (Final visit)
Population: The analysis population consisted of all participants who met all inclusion criteria, including a score of at least 13 on the CNS-LS, who received at least 1 dose of study drug, and who had at least 1 post-baseline efficacy measurement with QOL-VAS.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 298 | 108 | 103 | 87
Units on a scale | -3.13 (3.21) | -3.20 (2.98) | -2.66 (3.35) | -3.67 (3.29)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 2: Comparison: Dementia; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 3: Comparison: Stroke; Test type: Superiority or Other; p < 0.0001, One-sample t-test
Statistical Analysis 4: Comparison: Traumatic Brain Injury; Test type: Superiority or Other; p < 0.0001, One-sample t-test

9. Secondary Outcome: Percentage of Participants With Clinical Global Impression-Change (CGI-C) Score at Day 90
Description: CGI-C, an investigator-assessed scale was used to measure the overall treatment response. CGI-C, a 7-point (1-7) scale was rated as: very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse. Data is presented as percentage of participants with CGI-C score at Day 90. Percentages within a measure may not sum to 100.0 due to rounding. Percentages use the count of participants with non-missing data as the denominator.
Time Frame: Day 90 (Final visit)
Population: The analysis population consisted of all participants who met all inclusion criteria, including a score of at least 13 on the CNS-LS, who received at least 1 dose of study drug, and who had at least 1 post-baseline efficacy measurement with CGI-C.
Measure: Number; unit: Percentage of participants
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 261 | 102 | 91 | 68
Percentage of participants
  Very much improved | 33.7 | 30.4 | 33.0 | 39.7
  Much improved | 42.9 | 47.1 | 41.8 | 38.2
  Minimally improved | 13.4 | 13.7 | 14.3 | 11.8
  No change | 8.8 | 8.8 | 7.7 | 10.3
  Minimally worse | 0.8 | 0.0 | 2.2 | 0.0
  Much worse | 0.4 | 0.0 | 1.1 | 0.0
  Veru much worse | 0.0 | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Percentage of Participants With Patient Global Impression-Change (PGI-C) Score at Day 90
Description: PGI-C, a participant/participant's caregiver-assessed scale was used to measure participant overall treatment response. PGI-C, a 7-point (1-7) scale was rated as: very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse. Data is presented as percentage of participants with PGI-C score at Day 90. Percentages within a measure may not sum to 100.0 due to rounding. Percentages use the count of participants with non-missing data as the denominator.
Time Frame: Day 90 (Final visit)
Population: The analysis population consisted of all participants who met all inclusion criteria, including a score of at least 13 on the CNS-LS, who received at least 1 dose of study drug, and who had at least 1 post-baseline efficacy measurement with PGI-C.
Measure: Number; unit: Percentage of participants
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 261 | 102 | 92 | 67
Percentage of participants
  Very much improved | 32.6 | 28.4 | 33.7 | 37.3
  Much improved | 39.8 | 48.0 | 33.7 | 35.8
  Minimally improved | 18.8 | 14.7 | 21.7 | 20.9
  No change | 8.0 | 7.8 | 10.9 | 4.5
  Minimally worse | 0.4 | 1.0 | 0.0 | 0.0
  Much worse | 0.4 | 0.0 | 0.0 | 1.5
  Veru much worse | 0.0 | 0.0 | 0.0 | 0.0

11. Secondary Outcome: Percentage of Participants With Treatment Satisfaction Survey
Description: The treatment satisfaction survey was a 5 point single question survey that was administered by the site staff to the participant/participant's caregiver. Participants were asked to rate their response to treatment satisfaction as: very dissatisfied, somewhat dissatisfied, neither satisfied nor dissatisfied, somewhat satisfied, and very satisfied. Data is presented as percentage of participants with treatment satisfaction at Day 90. Percentages within a measure may not sum to 100.0 due to rounding. Percentages use the count of participants with non-missing data as the denominator.
Time Frame: Day 90 (Final visit)
Population: The mITT Population consisted of all participants who met all inclusion criteria, including a score of at least 13 on the CNS-LS, who received at least 1 dose of study drug, and who had at least 1 post-baseline efficacy measurement with CNS-LS.
Measure: Number; unit: Percentage of participants
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 261 | 102 | 92 | 67
Percentage of participants
  Very dissatisfied | 7.7 | 4.9 | 12.0 | 6.0
  Somewhat dissatisfied | 5.4 | 6.9 | 5.4 | 3.0
  Neither satisfied nor dissatisfied | 11.5 | 13.7 | 8.7 | 11.9
  Somewhat satisfied | 28.0 | 21.6 | 31.5 | 32.8
  Very satisfied | 47.5 | 52.9 | 42.4 | 46.3

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs (defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product) and SAEs (defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening [ie, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death], required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was as a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug) were assessed during the study.
Time Frame: From signing of informed consent up to 30 days after receiving the last dose of study drug or up to approximately 120 days
Population: The analysis was performed using the safety population that consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Number analyzed (Participants) | 367 | 134 | 113 | 120
Participants
  AEs | 132 | 49 | 40 | 43
  SAEs | 23 | 14 | 5 | 4

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 30 days after receiving the last dose of study drug or up to approximately 120 days
Arm/Group | Overall | Dementia | Stroke | Traumatic Brain Injury
Serious Adverse Events (participants affected / at risk) | 23/367 | 14/134 | 5/113 | 4/120
Other Adverse Events (participants affected / at risk) | 35/367 | 15/134 | 9/113 | 11/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=367) | Dementia (N=134) | Stroke (N=113) | Traumatic Brain Injury (N=120)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=367) | Dementia (N=134) | Stroke (N=113) | Traumatic Brain Injury (N=120)
Diarrhoea (Gastrointestinal disorders) | 20 | 5 | 5 | 10
Headache (Nervous system disorders) | 15 | 10 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other